CLINICAL TRIAL: NCT01003730
Title: The Effects of Different Ventilator Strategies on Inflammation and Injury in Normal Lungs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left the UMDNJ but may resume the study in her new place of employment.
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0120080132
Record Dates: First submitted 2009-10-21; First posted 2009-10-29 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Intraoperative protective ventilation strategies
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): High tidal volume (15mL/kg PBW0 with low PEEP (3cm H2O
  Interventions: Other: Ventilator settings
- 2 (Active Comparator): Low tidal volume (6mL/kg PBW) and high PEEP (3cm H2O)
  Interventions: Other: Ventilator settings
- 3 (Active Comparator): low tidal volume (6mL/kg PBW) and high PEEP (10cm H2O)
  Interventions: Other: Ventilator settings

INTERVENTIONS:
Other: Ventilator settings — Active Comparison of three different parameters of ventilator settings. Results of arterial blood gases and cytokine levels.

SUMMARY:
This research is being done to determine if there is a way the investigators can improve the techniques that they use to assist patients with their breathing during surgery. The majority of surgeries require patients to concurrently undergo general anesthesia. This usually includes a breathing tube and a machine that breathes for the patient during the duration of the surgery. The doctors would like to investigate the effects of this type of anesthesia to healthy adult patients and whether they can improve the way they give general anesthesia to patients. The investigators plan to ask approximately 200 patients to participate. If the patients decide to participate in the study,some additions will be made to the standard anesthetic care they receive. The patients will additionally be monitored for adequate oxygenation in their blood as well as level of inflammation in their blood and lungs. The patients' breathing tube will be bathed with warm normal saline and suctioned twice during the operation. When these procedures are done the patients will be asleep and not be aware of what is happening.

DETAILED DESCRIPTION:
The ability to provide mechanical ventilation that will not injure and may protect normal lungs during major surgical procedures of long duration may improve postoperative outcomes and decrease morbidity and mortality. The aim of the current study was to identify ventilator strategies that are less damaging to normal lungs. The investigators plan to compare three ventilation strategies commonly utilized in the operating room in normal lungs. One group will be ventilated with high tidal volume (15 mL/kg PBW) and low PEEP (3 cm H2O), another group ventilated with low tidal volume (6 mL/kg PBW) and low PEEP (3 cm H2O) and the final group ventilated with low tidal volume (6 mL/kg PBW) and high PEEP (10 cm H2O). This study will show the effects of these commonly used methods of ventilation on pulmonary mechanics, systemic and pulmonary inflammatory markers and outcomes in patients with normal lungs undergoing surgery of long duration.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery under general anesthesia expected to take 4 hours or more positioned supine for surgery

Exclusion Criteria:

* Subjects who have HIV or who have had Radiation or chemotherapy for cancer
* Subjects undergoing surgery on chest or lings
* Subjects who have obstructive sleep apnea (OSA), asthma, tuberculosis, chronic obstructive pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
cytokine levels in serum and bronchial aspirate | during the operative procedure

SECONDARY OUTCOMES:
arterial blood gases | during the operative procedure
subject post-operative outcome:mortality, pulmonary complications, major cardiac morbidity, LOS, readmission | wothin 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ellise Delphin, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ/University Hospital, Newark, New Jersey, United States

REFERENCES:
- [Background] Wrigge H, Zinserling J, Stuber F, von Spiegel T, Hering R, Wetegrove S, Hoeft A, Putensen C. Effects of mechanical ventilation on release of cytokines into systemic circulation in patients with normal pulmonary function. Anesthesiology. 2000 Dec;93(6):1413-7. doi: 10.1097/00000542-200012000-00012. PMID 11149435
- [Background] Wrigge H, Uhlig U, Baumgarten G, Menzenbach J, Zinserling J, Ernst M, Dromann D, Welz A, Uhlig S, Putensen C. Mechanical ventilation strategies and inflammatory responses to cardiac surgery: a prospective randomized clinical trial. Intensive Care Med. 2005 Oct;31(10):1379-87. doi: 10.1007/s00134-005-2767-1. Epub 2005 Aug 17. PMID 16132888